CLINICAL TRIAL: NCT05085509
Title: Foreign Body Removal With the Assistance of Ultrasound Guidance and Methylene Blue Staining
Brief Title: Foreign Body Removal With the Assistance of Ultrasound Guidance and Methylene Blue Staining in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuxi Su (Other)
Responsible Party: Sponsor-Investigator, Yuxi Su, Orthopaedic Department, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQMU-20210016
Record Dates: First submitted 2021-10-06; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Foreign Bodies; Ultrasound
MeSH Terms: conditions — Foreign Bodies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound (Experimental): Ultrasound guidance and methylene blue staining
  Interventions: Procedure: US guidance and MB staining
- Open surgery (Active Comparator): Open surgery without ultrasound guidance and methylene blue staining
  Interventions: Procedure: US guidance and MB staining

INTERVENTIONS:
Procedure: US guidance and MB staining — Ultrasound guidance and methylene blue staining

SUMMARY:
Soft-tissue foreign bodies (FB) are very commonly observed in pediatric emergency departments. Some are metallic and can be diagnosed easily via X-ray radiography, whereas others are radiolucent and are hence less easily diagnosed. Not all FB can be removed effectively, even via open surgery and C-arm guidance. This deficiency may potentially be addressed through the ultrasound (US) skills instrument, which is increasingly popular and is convenient for use in the operation room. In the current study, we evaluated the efficiency of FB removal with the assistance of US and methylene blue (MB) staining.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with soft-tissue foreign body
* Must have complete clinical data

Exclusion Criteria:

* Had other injuries
* Presented with more than 3 pieces foreign bodies

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Surgery time | Surgery end time
  Time from incision made to incision closure

SECONDARY OUTCOMES:
Blood loss | Surgery end time
  The blood loss of all the surgery time

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Foreign body removal with the assistance of ultrasound guidance and methylene blue staining in children